CLINICAL TRIAL: NCT00680797
Title: Metabolic Effects of Androgenicity in Aging Men and Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ARCD-034-04F
Record Dates: First submitted 2008-05-08; First posted 2008-05-20 (Estimated); Results first posted 2016-03-21 (Estimated); Last update posted 2017-06-15 (Actual); Status verified 2017-05

CONDITIONS: Aging; Insulin Resistance
Keywords: Aging; Hormones; Insulin resistance
MeSH Terms: conditions — Insulin Resistance | interventions — Testosterone; Estrogens

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- +T +E (Experimental): +Testosterone, +Estrogen
  Interventions: Drug: Testosterone; Drug: Estrogen
- +T -E (Experimental): +Testosterone, -Estrogen
  Interventions: Drug: Testosterone
- -T +E (Experimental): -Testosterone, +Estrogen
  Interventions: Drug: Estrogen
- -T -E (No Intervention): -Testosterone, -Estrogen

INTERVENTIONS:
Drug: Testosterone — Testosterone gel
  Arms: +T +E; +T -E
Drug: Estrogen — Estrogen patch
  Arms: +T +E; -T +E

SUMMARY:
The goal of this research study is to study the effect of testosterone or estrogen on blood sugar control and fat metabolism. Changes in hormone levels with age may affect risk factors for heart disease such as diabetes. Diabetes is a glandular condition associated with lack of the hormone insulin or an insensitivity to it resulting in problems with blood sugar control and fat metabolism. The effect of commonly used hormonal supplements such as testosterone by older adults on insulin and body composition is not well understood. In this study, the role of testosterone and estrogen on your ability to control blood sugar and your body composition will be assessed.

The investigators plan to study 60 subjects. All of these subjects will be healthy older men between the ages of 60-85 years old who are not on testosterone therapy. Subjects that are screened who have any clinically significant abnormalities detected on their screening physical exam or laboratory testing (e.g. Prostate Specific Antigen > 4), who have a history of prostate cancer, polycythemia, or who cannot take testosterone will not be included.

If a subject is eligible to participate after initial screening, that subject will take medications to adjust their hormone levels and have tests performed that measure insulin sensitivity and adiposity before and after these hormone medications. The outcomes that will be measured are: 1) insulin sensitivity, 2) hormone levels (total and free testosterone levels, sex hormone-binding globulin levels) and 3) body composition and abdominal adiposity.

ELIGIBILITY:
Inclusion Criteria:

* males age 60-85 years
* non-diabetic fasting glucose and 2-hour oral glucose tolerance test (OGTT)
* overall good general medical health and signed informed consent
* willing to travel to West Los Angeles VA and University of California, Los Angeles in Los Angeles, California

Exclusion Criteria:

* any clinically significant abnormalities detected on screening physical exam or laboratory testing (e.g. prostate specific antigen > 4)
* or other symptom or history of a significant underlying medical or psychiatric illness
* BMI < 20 or > 40
* subjects already on testosterone therapy or medications that might influence glucose regulation or hormone levels
* subjects with a history of deep venous thromboses, pulmonary embolism, breast cancer, prostate cancer, polycythemia or other contraindications to estrogen or testosterone

Ages: 60 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 33 (Actual)
Dates: Start 2005-01-01 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cathy C Lee, PhD, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (1):
- VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment methods included flyers and advertisement in local newspapers. Healthy Veteran and community participants who responded to to advertisement were screened by telephone for exclusion criteria. If no exclusion criteria were reported, participants were scheduled for a screening history and physical.
Period: Overall Study
Arm/Group | +T +E | +T -E | -T +E | -T -E
Started | 9 | 8 | 8 | 8
Completed | 9 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | +T +E | +T -E | -T +E | -T -E | Total
Number analyzed (Participants) | 9 | 8 | 8 | 8 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 3 | 2 | 4 | 14
  >=65 years | 4 | 5 | 6 | 4 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (8) | 66 (5) | 69 (6) | 63 (3) | 66 (6)
Sex/Gender, Customized [Number; unit: participants]
  Male | 9 | 8 | 8 | 8 | 33
Region of Enrollment [Number; unit: participants]
  United States | 9 | 8 | 8 | 8 | 33
Body-Mass-Index [Mean (Standard Deviation); unit: kilogram/meter squared] | 27.1 (4.9) | 28.6 (4.3) | 28.2 (4.1) | 29.0 (2.9) | 28.2 (4)
Total testosterone [Mean (Standard Deviation); unit: nanogram/deciliter] | 419.6 (146.5) | 418.9 (207.7) | 480.0 (231.7) | 558.3 (362.9) | 467.7 (242)

OUTCOME MEASURES:

1. Primary Outcome: Insulin Sensitivity
Description: As measured by change in insulin levels pre- and post-hormone changes
Time Frame: 6 weeks
Population: Two participants had missing values post-intervention therefore number of participants analyzed total 31.
Measure: Mean (Standard Deviation); unit: micro International Units/mL
Arm/Group | +T +E | +T -E | -T +E | -T -E
Number analyzed (Participants) | 8 | 8 | 8 | 7
micro International Units/mL | -0.16 (10.8) | 2.62 (5.47) | -0.50 (2.54) | 1.83 (4.24)
Statistical Analysis 1: Comparison: -T +E vs -T -E; The major outcome variable being presented is changes in insulin levels. Changes in insulin levels were analyzed using an ANCOVA model that adjusted for baseline insulin and age; Test type: Superiority or Other; p = 0.023, ANCOVA — Comparison of pre- to post-intervention insulin levels between the groups receiving E only versus the group receiving no hormone replacement
Statistical Analysis 2: Comparison: +T +E vs -T +E; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.042, ANCOVA — Comparison in the change in insulin levels between the groups receiving E with or without T

ADVERSE EVENTS:
Arm/Group | +T +E | +T -E | -T +E | -T -E
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/9 | 0/8 | 0/8 | 0/8

LIMITATIONS AND CAVEATS:
Small sample size may limit generalizability of these results. Follow-up studies are being conducted to further evaluate these results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No